CLINICAL TRIAL: NCT01227226
Title: Tear Osmolarity Over Time With Artificial Tears
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hom, Milton M., OD, FAAO (Individual)
Collaborators: Allergan (Industry)
Responsible Party: Milton M. Hom, OD, FAAO., Private Practice
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 06
Record Dates: First submitted 2010-10-21; First posted 2010-10-25 (Estimated); Last update posted 2011-02-07 (Estimated); Status verified 2011-02

CONDITIONS: Dry Eye
Keywords: Dry eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Refresh tears (Active Comparator): Allergan's Refresh tears artificial tear
  Interventions: Drug: Artificial tears
- Systane Ultra (Active Comparator): Alcon's Systane Ultra artificial tear
  Interventions: Drug: Artificial tears
- Visine (Active Comparator): Visine artificial tear
  Interventions: Drug: Artificial tears
- Blink tears (Active Comparator): AMO's blink tears artificial tear
  Interventions: Drug: Artificial tears

INTERVENTIONS:
Drug: Artificial tears — Instill one drop of artificial tears
  Other Names: Allergan's Refresh tears, Alcon's Systane Ultra, Johnson and Johnson's Visine, AMO's blink tears

SUMMARY:
The effect of artificial tears on tear osmolarity

DETAILED DESCRIPTION:
Tear osmolarity measures the amount of solutes in the human tear film. The higher the reading, the more likely the patient has dry eyes. Some say it has "potential to be the gold standard" of dry eye testing. The investigators study the tear osmolarity at different time points after instillation of artificial tears.

ELIGIBILITY:
Inclusion Criteria:

Between the ages of 18 and over inclusive. Males or females Any race or ethnic background Patient is in generally good & stable overall health. Patient likely to comply with study guidelines & study visits. Informed consent signed. Subjective evaluation of symptom of dryness (SESoD): Score 2 (Mild)

-

Exclusion Criteria:

Corneal refractive surgery within 6 months of this study. Intra-ocular surgery within 6 months or ocular laser surgery within 6 months. Pregnant or lactating women. Ocular pathology (includes glaucoma and cataract), which could impact results and/or place patient at risk.

Corneal staining Grade 3 or higher No Restasis for past 3 months Discontinue topical medications for at least 1 week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Tear osmolarity | 2 days
  Tear osmolarity measured with TearLab instrument

CONTACTS AND LOCATIONS:
Overall Officials: Milton M Hom, OD FAAO, Principal Investigator — Private Practice
Locations (1):
- Milton M. Hom, OD, FAAO., Azusa, California, United States